CLINICAL TRIAL: NCT02157740
Title: Assessment of Teleconsulting in Nursing Homes
Acronym: EVLINE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: TLM-EVLINE
Record Dates: First submitted 2014-05-27; First posted 2014-06-06 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Functionally-Impaired Elderly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control group before telemedicine: Residents of nursing homes without telemedicine before implementation of telemedicine in nursing homes with telemedicine
- Control group after telemedicine: Residents of nursing homes without telemedicine after implementation of telemedicine in nursing homes with telemedicine
- Exposed group, before telemedicine: Residents of nursing homes with telemedicine prior implementation of telemedicine
- Exposed group, after telemedicine: Residents of nursing homes with telemedicine after implementation of telemedicine
  Interventions: Device: Residents of nursing homes with telemedicine after implementation of telemedicine

INTERVENTIONS:
Device: Residents of nursing homes with telemedicine after implementation of telemedicine
  Groups: Exposed group, after telemedicine

SUMMARY:
The purpose of this study is to determine whether teleconsulting would be effective and cost-effective by reducing the patients transportations and the use of emergency units for nursing home residents requiring emergent or elective care.

ELIGIBILITY:
Inclusion Criteria:

* All residents of selected nursing homes

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nursing home residents
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Patient transportation to a emergency unit | Within 1 year after start of the study

SECONDARY OUTCOMES:
Transportation of the patient for a consultation | Within 1 year after start of the study
Mean length of hospital stay | Within 1 year after start of the study
Number of hospitalizations | Within 1 year after start of the study
Overall costs | Within 1 year after start of the study

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Durand-Zaleski, MD, PhD, Principal Investigator — DRCD URC Eco. Assistance Publique, Hôpitaux de Paris
Locations (9):
- France (9):
  - Résidence Le Sequoia, Châtenay-Malabry
  - Résidence Val de France, Domont
  - Résidence la Chanterelle, Le Pré-Saint-Gervais
  - Résidence les Noues, Montereau-Fault-Yonne
  - Résidence La Cerisaie, Poigny-la-Forêt
  - Résidence Saint Rémy, Saint Rémy Les Chevreuse
  - Résidence du Vexin, Saint-Clair-sur-Epte
  - Résidence Klarene, Tournan-en-Brie
  - Résidence Les Pastoureaux, Valenton

REFERENCES:
- [Background] Kidholm K, Ekeland AG, Jensen LK, Rasmussen J, Pedersen CD, Bowes A, Flottorp SA, Bech M. A model for assessment of telemedicine applications: mast. Int J Technol Assess Health Care. 2012 Jan;28(1):44-51. doi: 10.1017/S0266462311000638. PMID 22617736
- [Derived] Charrier N, Zarca K, Durand-Zaleski I, Calinaud C; ARS Ile de France telemedicine group. Efficacy and cost effectiveness of telemedicine for improving access to care in the Paris region: study protocols for eight trials. BMC Health Serv Res. 2016 Feb 8;16:45. doi: 10.1186/s12913-016-1281-1. PMID 26857558